CLINICAL TRIAL: NCT03504995
Title: Efficacy and Safety Assessment of Nanoknife (AngyoDynamics, USA) for Irreversible Electroporation (IRE) of Localized Prostate Cancer.
Brief Title: Efficacy and Safety Assessment of IRE of Localized Prostate Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Science of RI of Uronephrology and Reproductive Health, I.M. Sechenov First Moscow State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sechenov-IRE18
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: Prostate; Irreversible Electroporation; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- IRE patients (Experimental): patients who will underwent 'Focal irreversible electroporation of the prostate cancer'
  Interventions: Device: Focal irreversible electroporation of the prostate cancer

INTERVENTIONS:
Device: Focal irreversible electroporation of the prostate cancer — Irreversible electroporation is a non-thermal tissue ablation technique in which short duration electrical fields are used to permanently permeabilize the cell membrane.

SUMMARY:
The purpose of this study is to evaluate safety and short-term oncological efficacy of the NanoKnife Irreversible Electroporation System for localised prostate cancer.

Irreversible electroporation (IRE) is the method of focal treatment for prostate cancer, which is already proven by FDA as method of the surgical ablation of soft tissue. It has not received clearance for the therapy or treatment of any specific disease or condition.

DETAILED DESCRIPTION:
Irreversible electroporation is a newly developed non-thermal tissue ablation technique in which short duration electrical fields are used to form permanent nanoscale defects in the cell membrane which leads to cell apoptosis. Thus, IRE is a non-thermal technique, which means that changes associated with tissue freezing or heating are not relevant.

Moreover, animal studies of IRE in the canine prostate have demonstrated that structures such as ejaculatory ducts, neurovascular bundles, blood vessels, and the urethra heal normally after ablation. The reason is that collagen matrix during treatment with IRE is not destroyed thus allowing for a large structures (blood vessels, nerves, etc.) to heal normally.

This study is a prospective and non-randomized with one group of 10 patients eligible for focal therapy of prostate cancer with IRE (eligibility defined by this protocol).

Before the surgery all patients will underwent transperineal MRI-fusion biopsy to localize the prostate cancer foci.

Objectives of the study: to asses safety of IRE in patients with localized PCa, to asses short-term oncologic efficacy of IRE in patients with localized PCa, to asses functional outcomes after IRE.

All patients will be followed up for 1 year (each 3 months).

ELIGIBILITY:
Inclusion Criteria:

* Verified with MR-fusion biopsy localized Pca
* PSA < 15 ng/ml
* Gleason score 3+3=6; 3+4=7 OR Grade Group 1 and 2
* Life expectancy > 10 years
* No post-void residual urine or infravesical obstruction

Exclusion Criteria:

* patients with artificial cardiac pacemaker
* patients without rectum
* patients not eligible for general anesthesia
* PIRADS<3
* patients after primary Pca treatment
* hormonal therapy six months before the study
* radiotherapy of pelvic organs
* urinary infection
* extracapsular Pca
* patients with metastatic lesions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
PSA level | 3 months, 6 months, 9 months, 12 months.
  Stable decrese of PSA level after surgery (<1 ng/ml)
Complications | 1 year
  Short and long term surgical complications

SECONDARY OUTCOMES:
IPSS (International Prostate Symptom Score, range from 5 to 30) | 1 year
  International Prostate Symptom Score
QoL (Quality of Life score, range 1-6) | 1 year
  Quality of Life Score
Qmax | 1 year
  Maximal urine flow rate
IIEF | 1 year
  International Index of Erectile Function - Erectile function assessment (range 1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Enikeev, MD, PhD, Study Director — I.M. Sechenov First Moscow State Medcal University
Locations (1):
- Clinic of Urology, Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rubinsky B. Irreversible electroporation in medicine. Technol Cancer Res Treat. 2007 Aug;6(4):255-60. doi: 10.1177/153303460700600401. PMID 17668932
- [Background] Scheltema MJ, Chang JI, Bohm M, van den Bos W, Blazevski A, Gielchinsky I, Kalsbeek AMF, van Leeuwen PJ, Nguyen TV, de Reijke TM, Siriwardana AR, Thompson JE, de la Rosette JJ, Stricker PD. Pair-matched patient-reported quality of life and early oncological control following focal irreversible electroporation versus robot-assisted radical prostatectomy. World J Urol. 2018 Sep;36(9):1383-1389. doi: 10.1007/s00345-018-2281-z. Epub 2018 Mar 28. PMID 29594551